CLINICAL TRIAL: NCT02577419
Title: Optimizing Growth in Infants Receiving Modified Fat Breast Milk for the Treatment of Chylothorax Following Cardiothoracic Surgery
Brief Title: Optimizing Growth in Infants Receiving Modified Fat Breast Milk for the Treatment of Chylothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Labatt Family Heart Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, Physiology and Experimental Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000048134
Record Dates: First submitted 2015-10-01; First posted 2015-10-16 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Chylothorax
Keywords: breast milk; chylothorax; infants; cardiac surgery; modified fat breast milk
MeSH Terms: conditions — Chylothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Target Fortification (Experimental)
  Interventions: Other: Target Fortification
- Higher Initial Concentration (Experimental)
  Interventions: Other: Higher Initial Concentration
- Portagen Growth Reference (Active Comparator)
  Interventions: Other: Portagen Formula

INTERVENTIONS:
Other: Target Fortification
  Arms: Target Fortification
Other: Higher Initial Concentration
  Arms: Higher Initial Concentration
Other: Portagen Formula
  Arms: Portagen Growth Reference

SUMMARY:
Breast milk is the reference normative standard for infant feeding. When an infant is diagnosed with chylothorax, provision of breast milk must be temporarily discontinued due to the presence of long chain triglycerides (LCT) that contribute to persistent chylous drainage. In its place, the infant is prescribed a therapeutic formula high in medium chain triglycerides (MCT) as treatment for chylothorax. Families and health care providers are interested in using breast milk, in a modified fat form, as treatment for chylothorax instead. This study will assess growth in infants receiving one of two nutrient enriched modified fat breast milk (MFBM) treatments for chylothorax. If either of the proposed nutrient enrichment methods support growth, MFBM will become a standard chylothorax treatment option for infants at SickKids.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of chylothorax following cardiothoracic surgery
* previously receiving a minimum of 50% of feeds from breast milk 3 days prior to surgical procedure
* parents/caregivers would like to continue to provide breast milk during chylothorax treatment

Exclusion Criteria:

* diagnoses of chylothorax classified as either congenital, obstructive, or traumatic not following cardiothoracic surgery
* patient has a chromosomal anomaly that affects growth (i.e. Trisomy 21, Trisomy 18 etc.)
* patient receiving less than 50% of feeds from breast milk (or mother does not have intention to provide breast milk)
* neither parent/caregiver/family member able to communicate effectively in English

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Growth - weight | Throughout chylothorax treatment (average 6 weeks); daily in hospital; weekly as outpatient
  z-score for weight-for-age
Growth - length | Throughout chylothorax treatment (average 6 weeks); calculated daily in hospital; weekly as outpatient
  z-score for length-for-age
Growth - head circumference | Throughout chylothorax treatment (average 6 weeks); calculated daily in hospital; weekly as outpatient
  z-score for head circumference-for-age

SECONDARY OUTCOMES:
Feed volume intakes | Throughout chylothorax treatment (average 6 weeks); calculated daily in hospital; weekly as outpatient
Energy intakes | Throughout chylothorax treatment (average 6 weeks); calculated daily in hospital; weekly as outpatient
Protein intakes | Throughout chylothorax treatment (average 6 weeks); calculated daily in hospital; weekly as outpatient
Solid food intakes (type, grams at home measured using a scale (CS2000; Ohaus)) | Throughout chylothorax treatment (average 6 weeks); daily in hospital; weekly as outpatient
Volume of chest tube drainage | Throughout chylothorax treatment (average 6 weeks); daily in hospital
  ml/kg/day
Duration of chest tube drainage | Throughout chylothorax treatment (average 6 weeks); daily in hospital
  measured in post-operative days
Morbidities - hospital re-admission(s) | Throughout chylothorax treatment (average 6 weeks)
Morbidities - reaccumulation of chylous fluid | Throughout chylothorax treatment (average 6 weeks)
Morbidities - prevalence of serious adverse events | Throughout chylothorax treatment (average 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD RD, Principal Investigator — The Hospital for Sick Children; Sara DiLauro, MSc(c) RD, Principal Investigator — The Hospital for Sick Children; Jennifer Russell, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kocel SL, Russell J, O'Connor DL. Fat-Modified Breast Milk Resolves Chylous Pleural Effusion in Infants With Postsurgical Chylothorax but Is Associated With Slow Growth. JPEN J Parenter Enteral Nutr. 2016 May;40(4):543-51. doi: 10.1177/0148607114566464. Epub 2015 Jan 5. PMID 25560680
- [Background] DiLauro S, Russell J, McCrindle BW, Tomlinson C, Unger S, O'Connor DL. Growth of cardiac infants with post-surgical chylothorax can be supported using modified fat breast milk with proactive nutrient-enrichment and advancement feeding protocols; an open-label trial. Clin Nutr ESPEN. 2020 Aug;38:19-27. doi: 10.1016/j.clnesp.2020.05.001. Epub 2020 May 23. PMID 32690156